CLINICAL TRIAL: NCT02638506
Title: Randomized Controlled Trial Evaluating the Additive Value of Intranasal Fentanyl on Ibuprofen in the Pain Management of Children With Moderate to Severe Headaches
Brief Title: RCT Evaluating Intranasal Fentanyl in the Pain Management of Children With Headaches
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Covid restrictions
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Serge Gouin, Associate Professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INF2016-1028
Record Dates: First submitted 2015-12-21; First posted 2015-12-23 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Headaches
Keywords: Headaches, Migraines, Fentanyl
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal Fentanyl (Experimental): All patients will receive a 1.5 mcg⁄kg dose of fentanyl or an equivalent volume of similar looking placebo. This will be administered intranasally via a mucosal atomiser device (MAD) using 50 mcg/mL solution with a 2 mL syringe.
  Interventions: Drug: Fentanyl
- Salinex (Placebo Comparator): All patients will receive a 1.5 mcg⁄kg dose of fentanyl or an equivalent volume of similar looking placebo. This will be administered intranasally via a mucosal atomiser device (MAD) using 50 mcg/mL solution with a 2 mL syringe.
  Interventions: Other: Salinex

INTERVENTIONS:
Drug: Fentanyl — All patients will receive a 1.5 mcg⁄kg dose of fentanyl. This will be administered intranasally via a mucosal atomiser device (MAD) using 50 mcg/mL solution with a 2 mL syringe
  Other Names: Fentanyl citrate
  Arms: Intranasal Fentanyl
Other: Salinex — All patients will receive an equivalent volume of similar looking placebo to fentanyl (1.5 mcg/kg dose). This will be administered intranasally via a mucosal atomiser device (MAD) using 50 mcg/mL solution with a 2 mL syringe
  Arms: Salinex

SUMMARY:
Background : Headaches are a common presentation for children consulting to the Emergency Department (ED). However, only few studies have evaluated the rapid pain improvement provided by medications in the acute management of headaches in the pediatric population.

Objective : To evaluate pain reduction provided by intranasal fentanyl (INF) compared to placebo in addition to ibuprofen for children presenting to a pediatric ED with moderate to severe headaches.

Methods : A single-center, double-blind, randomized, placebo controlled clinical trial will be conducted in an urban, university-affiliated, tertiary care pediatric hospital ED. All children eight to 18 years old who will present to the ED with headaches as a main chief complaint and with pain of ≥ 36 mm out of 100 on Visual Analog Scale (VAS) will be recruited. Study participants will be randomly allocated to receive INF 1.5 mcg/kg (maximum dose of 100 mcg) or similar volume of a placebo solution via an atomizer. Co-administration of oral ibuprofen 10 mg/kg (maximum dose of 600 mg) will also be provided to the two groups if not received in the previous 4 hours. The primary outcome will be the mean pain rating reduction at 15 minutes. The secondary outcomes will be mean pain reduction at 30 and 60 minutes, patient's and parental satisfaction levels, percent of being pain free, sedation score, immediate and within 72 hours adverse events, additional ED analgesics and other medications, length of ED stay, disposition outcomes, hospital admission rate and ED revisit rate within 72 hours. The primary analysis will use an intention-to-treat approach to compare mean pain score reduction between the two groups using a Student's T-test. The sample size of 60 participants per arm was calculated to have a power of 80% to identify a difference of 10 mm in the VAS.

Expected results : Our study might demonstrate that INF provides additional pain relief for children presenting to an ED with headaches. Providing INF could relieve their symptoms more quickly, potentially improve patient's and family's satisfaction, possibly reduce the length of their ED stay and consequently, have a significant impact on patient quality of care and cost-effectiveness.

DETAILED DESCRIPTION:
The primary objective of the present study would be to determine the additive value on analgesic effectiveness of INF in children aged eight to 18 years with acute moderate to severe headaches. We would also aim to gather information on the safety and acceptability of INF for headaches. We believe that providing INF for moderate to severe headaches will decrease pain levels in children aged 8 to 18 years old.

We will perform a prospective, double-blind, randomized placebo-controlled clinical trial.

The study setting will be a single center, urban, university-based, tertiary care pediatric university-affiliated hospital ED with an annual census of 75,000 patient visits. The study should be conducted between 2015-2018.

Study population : Inclusion criteria will consist of children aged eight to 18 years who present to the pediatric ED with a chief complaint of headaches, regardless of the type, with a moderate or severe pain score. Pain was considered at least moderate if superior or equal to 36 mm on the VAS as demonstrated by Hirschfeld et. Al. This level have been chosen because it has been recognized that adequate sensitivity in analgesia trials for acute pain can only be obtained if patients experience at least moderate pain before administration of any treatment.

Intervention: All patients will receive a 1.5 mcg⁄kg dose of fentanyl or an equivalent volume of similar looking placebo. This will be administered intranasally via a mucosal atomiser device (MAD) using 50 mcg/mL solution with a 2 mL syringe. Prior studies have shown that this dose is as effective as IV or IM morphine and provides a bioavailability which is 71% of the IV dose. The minimum dose prescribed will be 20 mcg, to ensure delivery of 15 mcg of fentanyl to a 10 kg child, allowing for the MAD dead space of 0.1 mL (5 mcg of fentanyl). For analgesic dose-volumes equal to and less than 0.5 mL, the entire dose will be administered in one nostril; doses above 0.5 mL will be divided equally and administered to both nostrils. Concentrated medications in a small volume (0.2-0.3 mL per nostril) are ideal, whereas volumes in excess of 1 mL per nostril are not reliably absorbed as a result of mucosal surface saturation and runoff from the nasal cavity. The maximum dose administered will be 100 mcg due to volume constraints. The placebo solution will consist of normal saline that would be delivered via the proposed atomiser. The value administered will be adjusted to the patients weight as for the active study medication. No additional dose of either study medication would be provided. A MAD have been chosen because it is suggested to increase the mucosal coverage and absorption of the medication by atomizing particles and decreasing the amount of medication lost due to swallowing.

Oral ibuprofen (10 mg/kg) (maximum dose of 600 mg) will also be administered within the first 15 minutes of intranasal administration of the study medication unless it had been given in the previous 4 hours. It has been chosen over acetaminophen because a direct comparison has shown that complete pain relief after two hours is achieved twice as frequently with ibuprofen.

The randomization process will occur at the local pharmacy and randomization allotment will be known only by a pharmacist who is not involved in the study. Therefore, all providers involved in the patient's care and patients will be blinded to group assignment until data analysis completion. The participant will be randomly assigned to one of the two groups as follows : 1) INF 1.5 mcg/kg and 2) placebo solution, given via an atomizer (MAD device: MAD Nasal, U.S. Patent #6,112,743, Wolfe-Tory Medical, Inc., 79 West 4500 South, Salt Lake City, Utah 84107).

The study medications will be provided to the ED by the local pharmacy. For each randomized patient, a consecutive study medication package will be opened in the ED. Each study package will contain a study medication (either generic fentanyl bottle or saline bottle), a syringe and an atomizer for delivery. An on-site nurse will withdraw the study medication from the specific bottle provided in the package and will deliver the study medication to the patient. The study research assistant will remain blinded. At the pharmacy, the patient's identification will be coded so that only a user having the access code will be able to identify participants.

Procedure : Every patient will be weighed in triage. Enrollment will be limited to times when a research assistant is available. A research assistant will recruit the patients after a pediatric ED physician has assessed them and once the symptoms of headaches are clearly established. The pain associated with headaches will be assessed by using the VAS, which has been validated for the use in children aged eight years and older across a variety of clinical settings and has an excellent interrater-reliability and validity in analgesia research.

Once eligibility and exclusion criteria will be confirmed, caregivers will be given written and verbal study information. Written consent for enrolment will be gained from both the accompanying parent and the child, when appropriate. The research assistant will use timers to coordinate all the events. At baseline, before any intervention, the VAS score, baseline vital signs and sedation score (UMSS) will be recorded by the research assistant. For the assessment of the VAS score, the children will be asked to mark on a standardized data collection booklet, the level of their pain on a 100-mm non hatched VAS scale with at one end "no pain" and at the other "worst pain ever" with the following, verbatim: "Show me on the line the level of your pain: here is no pain; there is the worst possible pain." The patient will then cross a line to indicate his or her level of pain. All measurements will be recorded to the closest 1 mm.

At time zero, the solution contained in a syringe will be administered by the on-site nurse to the anterior aspect of the participant's nasal cavity over few seconds. The dose (or half of it, if necessary) will be administered into one of the patient's nostrils with the MAD. The second half of the dose, if needed, will be administered in the contralateral nostril using the same MAD. Younger children will have the medication administered while sitting in the lap of a parent, with their heads reclined and necks hyperextended. Older children will receive the medication while lying in a semi recumbent position on the gurney. No additional dose would be provided. The research assistant will remain blinded to which medication the patient has received.

At the fifteenth, thirtieth and sixtieth minute post-intervention, the research assistant will obtain a pain score via the VAS from the patient and ask for the change in their pain. They will be asked to give a verbal rating of their pain as 'a lot less', 'a little less', 'the same', 'a little more' or 'a lot more' compared to the initial baseline, at time zero and reassess level of pain on the VAS as used previously. Children will not be permitted to refer to previous scales markings and will remain blinded to their prior scores. The sedation score will also be recorded using the University of Michigan Sedation Scale (UMSS) which overall validity was demonstrated and declared as a simple, valid and reliable tool that facilitates rapid and frequent assessment and documentation of depth of sedation in children. The vital signs will also be taken at these intervals.

A detailed demographic and clinical data will also be collected after the study medication administration. A standardized questionnaire of the patient's present and past headaches, will be completed by the research assistant during their stay in the pediatric ED. The questionnaire will include questions on duration, location, description of pain, associated symptoms of the present headache and past medical history.

No other meds, IV fluids, IV procedures or other painful procedures will be done during the study period unless the patient's condition changes or deteriorates. If any of these procedure is needed during the study period, the patient will be withdrawn from the study and will be treated according of his state of health.

At the sixtieth minute of the study, marking the end of the study, patients who had assented to the study and parents will be asked to rate their satisfaction on the efficacy of the study medication on a Likert scale ('strongly disagree' 'disagree', 'neither agree nor disagree', 'agree', or 'strongly agree'). This satisfaction scale will be given to patients and parents after the last pain score was obtained. The study would be then completed, and further care will be at the discretion of the attending pediatric ED medical staff.

A follow-up call by a research assistant will be done at 72 hours after discharge to assess headache recurrence, late medication side effects, and a return to another medical facility. All children hospitalized will also be reached.

A chart review will be done by a member of the research team to collect final pediatric ED diagnosis as well as any additional investigations (e.g. CT scan, consultation with a neurologist, blood tests, TSH, etc.).

Data will be collected using pediatric ED medical records of recruited patients and the sociodemographic questionnaire completed by a research assistant. The results of all other variables: VAS, UMSS and satisfaction score will be collected in real time by the research assistant during the pediatric ED stay.

A data collection form will be used, and these forms will be later cross-referenced with the patient's clinical records by a member of the research team to verify correct documentation and eligibility.

Sample size and statistics :

This is the first study evaluating pain related to all types of headaches in children. Accordingly, no previous study perfectly matches our design to infer sample size. However, two previous studies evaluated an intervention provided to decrease acute pain secondary to migraine in children using the VAS. These studies reported a standard deviation of 18.5 and 20 mm. Powell et al found the minimum clinically significant difference (MCSD) in VAS pain score for children aged 8 to 15 years (on a 100-mm VAS scale) to be 10 mm (95% confidence interval 7 to 12 mm). In studies of populations, differences of less than this amount, even if statistically significant, are unlikely to be of clinical significance. Previous research in adults has found the same MCSD in VAS pain scores and did not differ in adults with age, sex, or cause of pain. Based on these data, using an alpha value of 0,05 and a power of 80%, it was estimated that we need, 57 patients per group. Accounting to a maximal 5% drop-off rate, we inflated this number to 60 participants per group.

All data will be entered in an excel database (Microsoft Inc., Richmond, WA) and will be analyzed with SPSS v21 (IBM Inc). The primary study analysis will be a Student's T-test to compare the mean differences in scores between the intervention group and the placebo group. An intention-to-treat approach will be used. Also, secondary analyses will be performed using a Student's T-test for continuous variables and a Pearson Chi-square test for categorical variables. The 95% confidence intervals will be measured for each result.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria will consist of children aged eight to 18 years who present to the pediatric ED with a chief complaint of headaches, regardless of the type, with a moderate or severe pain score.

Pain was considered at least moderate if superior or equal to 36 mm on the VAS as demonstrated by Hirschfeld et. Al. This level have been chosen because it has been recognized that adequate sensitivity in analgesia trials for acute pain can only be obtained if patients experience at least moderate pain before administration of any treatment.

Exclusion Criteria:

* 1. Allergy or any contra-indication to opioids and-or ibuprofen 2. Previous participation in study to preserve the statistic independence of each participant 3. Caregiver unable to provide consent (language barrier or lack of caregiver presence) 4. Circumstance which, in the opinion of the investigator, would adversely affect their participation in the trial such as a medical or psychiatric condition or a language barrier (neither French or English) 5. Nasopharyngeal anomalies, blockage or traumatized preventing nasal administration 6. Suspicion of life-threatening illness such as acute intracranial haemorrhage, meningitis, encephalopathy, or intracranial cerebral vascular occlusion 7. Signs of intracranial pressure or suspicion of intracerebral process such as mass or tumors (altered mental status, focal neurological deficit, etc.) 8. Any head injury with possible associate intracranial injury in the past 14 daysRecent or acute head injury 9. Current opioid use or opioid antagonist use 10. Intoxication

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2016-01; Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the difference of the subjects' self-reported pain scores as assessed by the VAS at the fifteenth minute after administration of the initial drug therapy, which correspond to its peak analgesic effect. | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Serge Gouin, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Ste-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No